CLINICAL TRIAL: NCT02447302
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Study to Investigate the Safety and Efficacy of APD334 in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: Safety and Efficacy of Etrasimod (APD334) in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APD334-003; 2015-001942-28 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Etrasimod Low Dose (Experimental): Oral, low dose, daily for 12 Weeks
  Interventions: Drug: Etrasimod
- Etrasimod High Dose (Experimental): Oral, high dose, daily for 12 weeks
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator): Oral, placebo, daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod
  Other Names: APD334
  Arms: Etrasimod High Dose; Etrasimod Low Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether etrasimod is a safe and effective treatment for ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Moderately to severely active ulcerative colitis defined as a 3-component Mayo Clinic score
* Evidence of colonic ulcerative colitis activity on endoscopy

Exclusion Criteria:

* Within 30 days prior to randomization, receipt of any of the following for the treatment of underlying disease: Non-biologic therapies (eg, cyclosporine, tacrolimus, tofacitinib, thalidomide), a non-biologic investigational therapy or an approved non-biologic therapy in an investigational protocol
* Within 60 days prior to randomization, receipt of any of the following: Infliximab, adalimumab, golimumab, certolizumab, vedolizumab, any other investigational or approved biologic agent
* Any prior exposure to natalizumab, efalizumab, or rituximab

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (134):
- United States (30):
  - Arena 1119, Birmingham, Alabama
  - Arena 1133, Dothan, Alabama
  - Arena 1143, Thousand Oaks, California
  - Arena 1107, Hollywood, Florida
  - Arena 1138, Miami, Florida
  - Arena 1123, Naples, Florida
  - Arena 1141, Orlando, Florida
  - Arena 1106, Port Orange, Florida
  - Arena 1137, Sweetwater, Florida
  - Arena 1131, Chicago, Illinois
  - Arena 1139, Hoffman Estates, Illinois
  - Arena 1127, Urbana, Illinois
  - Arena 1142, Traverse City, Michigan
  - Arena 1111, Troy, Michigan
  - Arena 1109, Great Neck, New York
  - Arena 1114, Rochester, New York
  - Arena 1118, Raleigh, North Carolina
  - Arena 1112, Cincinnati, Ohio
  - Arena 1117, Pittsburgh, Pennsylvania
  - Arena 1105, Germantown, Tennessee
  - Arena 1102, Hermitage, Tennessee
  - Arena 1136, DeSoto, Texas
  - Arena 1121, Houston, Texas
  - Arena 1116, Temple, Texas
  - Arena 1103, Ogden, Utah
  - Arena 1130, Richmond, Virginia
  - Arena 1128, Roanoke, Virginia
  - Arena 1115, Seattle, Washington
  - Arena 1101, Seattle, Washington
  - Arena 1108, Wauwatosa, Wisconsin
- Australia (3):
  - Arena 1604, Kingswood
  - Arena 1605, Randwick
  - Arena 1607, Subiaco
- Arena 1490, Vienna, Austria
- Belgium (3):
  - Arena 1472, Edegem
  - Arena 1464, Kortrijk
  - Arena 1473, Leuven
- Bulgaria (6):
  - Arena 1421, Rousse
  - Arena 1409, Sofia
  - Arena 1410, Sofia
  - Arena 1417, Sofia
  - Arena 1407, Sofia
  - Arena 1425, Varna
- Canada (6):
  - Arena 1202, Winnipeg, Manitoba
  - Arena 1210, Bridgewater, Nova Scotia
  - Arena 1208, Greater Sudbury, Ontario
  - Arena 1209, Greater Sudbury, Ontario
  - Arena 1206, London, Ontario
  - Arena 1204, Toronto, Ontario
- Arena 1455, Prague, Czechia
- France (7):
  - Arena 1443, Amiens
  - Arena 1418, Clichy
  - Arena 1437, Lille
  - Arena 1476, Paris
  - Arena 1480, Pierre-Bénite
  - Arena 1423, Saint-Etienne
  - Arena 1457, Vandœuvre-lès-Nancy
- Germany (7):
  - Arena 1479, Hamburg
  - Arena 1422, Hamburg
  - Arena 1470, Hanover
  - Arena 1446, Kiel
  - Arena 1489, Leipzig
  - Arena 1497, Oldenburg
  - Arena 1444, Ulm
- Hungary (7):
  - Arena 1478, Békéscsaba
  - Arena 1471, Budapest
  - Arena 1492, Budapest
  - Arena 1431, Budapest
  - Arena 1505, Debrecen
  - Arena 1474, Debrecen
  - Arena 1477, Szombathely
- Israel (5):
  - Arena 1705, Beersheba
  - Arena 1702, Haifa
  - Arena 1706, Holon
  - Arena 1704, Jerusalem
  - Arena 1703, Petah Tikva
- Latvia (2):
  - Arena 1462, Riga
  - Arena 1475, Riga
- Arena 1484, Vilnius, Lithuania
- Arena 1601, Christchurch, New Zealand
- Poland (9):
  - Arena 1439, Bydgoszcz
  - Arena 1486, Elblag
  - Arena 1495, Kielce
  - Arena 1451, Krakow
  - Arena 1438, Lodz
  - Arena 1458, Poznan
  - Arena 1428, Rzeszów
  - Arena 1456, Sopot
  - Arena 1494, Wroclaw
- Romania (7):
  - Arena 1441, Bucharest
  - Arena 1491, Bucharest
  - Arena 1406, Bucharest
  - Arena 1436, Iași
  - Arena 1420, Oradea
  - Arena 1405, Timișoara
  - Arena 1493, Timișoara
- Russia (10):
  - Arena 1440, Kazan'
  - Arena 1500, Krasnoyarsk
  - Arena 1504, Novosibirsk
  - Arena 1419, Rostov-on-Don
  - Arena 1452, Ryazan
  - Arena 1498, Saint Petersburg
  - Arena 1467, Saint Petersburg
  - Arena 1448, Saint Petersburg
  - Arena 1447, Saint Petersburg
  - Arena 1465, Samara
- South Korea (7):
  - Arena 1613, Busan
  - Arena 1614, Daegu
  - Arena 1610, Incheon
  - Arena 1612, Seoul
  - Arena 1611, Seoul
  - Arena 1608, Suwon
  - Arena 1615, Wŏnju
- Spain (6):
  - Arena 1403, Barcelona
  - Arena 1460, Barcelona
  - Arena 1481, Madrid
  - Arena 1430, Pontevedra
  - Arena 1432, Santiago de Compostela
  - Arena 1469, Seville
- Ukraine (12):
  - Arena 1424, Chernivtsi
  - Arena 1445, Ivano-Frankivsk
  - Arena 1454, Kharkiv
  - Arena 1459, Kharkiv
  - Arena 1466, Kiev
  - Arena 1408, Kyiv
  - Arena 1502, Kyiv
  - Arena 1506, Kyiv
  - Arena 1414, Odesa
  - Arena 1433, Uzhhorod
  - Arena 1416, Vinnytsia
  - Arena 1501, Vinnytsia
- United Kingdom (3):
  - Arena 1302, London
  - Arena 1304, Torquay
  - Arena 1303, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermeire S, Rubin DT, Peyrin-Biroulet L, Dubinsky MC, Regueiro M, Irving PM, Goetsch M, Lazin K, Gu G, Wu J, Modesto I, McDonnell A, Guo X, Green J, Dalam AB, Yarur AJ. Cardiovascular events observed among patients in the etrasimod clinical programme: an integrated safety analysis of patients with moderately to severely active ulcerative colitis. BMJ Open Gastroenterol. 2025 Jan 8;12(1):e001516. doi: 10.1136/bmjgast-2024-001516. PMID 39778975
- [Derived] Lees CW, Torres J, Leung Y, Vermeire S, Fellmann M, Modesto I, McDonnell A, Lazin K, Keating M, Goetsch M, Wu J, Loftus EV Jr. Non-serious adverse events in patients with ulcerative colitis receiving etrasimod: an analysis of the phase II OASIS and phase III ELEVATE UC 52 and ELEVATE UC 12 clinical trials. Therap Adv Gastroenterol. 2024 Nov 7;17:17562848241293643. doi: 10.1177/17562848241293643. eCollection 2024. PMID 39526078
- [Derived] Yarur AJ, Chiorean MV, Panes J, Jairath V, Zhang J, Rabbat CJ, Sandborn WJ, Vermeire S, Peyrin-Biroulet L. Achievement of Clinical, Endoscopic, and Histological Outcomes in Patients with Ulcerative Colitis Treated with Etrasimod, and Association with Faecal Calprotectin and C-reactive Protein: Results From the Phase 2 OASIS Trial. J Crohns Colitis. 2024 Jun 3;18(6):885-894. doi: 10.1093/ecco-jcc/jjae007. PMID 38245818
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Zhang J, Chiorean M, Vermeire S, Lee SD, Kuhbacher T, Yacyshyn B, Cabell CH, Naik SU, Klassen P, Panes J. Efficacy and Safety of Etrasimod in a Phase 2 Randomized Trial of Patients With Ulcerative Colitis. Gastroenterology. 2020 Feb;158(3):550-561. doi: 10.1053/j.gastro.2019.10.035. Epub 2019 Nov 9. PMID 31711921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a screening period (up to 28 days), a double-blind induction treatment period (12 weeks), and a possible follow-up visit (2 weeks after the last study visit). The target population consisted of male or female participants aged between 18 and 80 years (inclusive), with moderately to severely active Ulcerative Colitis.
Pre-assignment Details: During the screening period (Days -28 to -1), participants were evaluated for study entry based on the inclusion and exclusion criteria. Screening procedures to evaluate participant eligibility for the study were to be conducted within 28 days prior to study drug administration on Day 1.
Groups:
- Etrasimod 1 mg: Etrasimod 1 mg was administered orally once daily for 12 weeks, administered with approximately 240 mL (8 ounces) of water. The study drug was to be taken on an empty stomach after an overnight fast of approximately 8 hours.
- Etrasimod 2 mg: Etrasimod 2 mg was administered orally once daily for 12 weeks, administered with approximately 240 mL (8 ounces) of water. The study drug was to be taken on an empty stomach after an overnight fast of approximately 8 hours.
- Placebo: Placebo was administered orally once daily for 12 weeks, administered with approximately 240 mL (8 ounces) of water. Placebo was to be taken on an empty stomach after an overnight fast of approximately 8 hours.
Period: Overall Study
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Started | 52 | 50 | 54
Completed | 47 | 46 | 48
Not Completed | 5 | 4 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Adverse Event | 4 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 5
Not completed — Sponsor Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed using the safety population that consisted of all randomized participants who received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo | Total
Number analyzed (Participants) | 52 | 50 | 54 | 156
Age, Continuous [Median (Full Range); unit: years] | 44.0 [21 to 64] | 38.5 [21 to 67] | 46.0 [20 to 73] | 42 [20 to 73]
Age, Customized [Number; unit: Subjects]
  Adults (18-64 years) | 52 | 49 | 49 | 150
  From 65-80 years | 0 | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 22 | 67
  Male | 30 | 27 | 32 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 7
  Not Hispanic or Latino | 49 | 49 | 51 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 47 | 49 | 51 | 147
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Adapted Mayo Score (MCS) [Mean (Standard Deviation); unit: score on a scale] — The adapted MCS was used to measure disease activity of ulcerative colitis. It consisted of 3 subscores (stool frequency, rectal bleeding, and findings of endoscopy), each of which was rated on a scale from 0 to 3, indicating normal to severe. The adapted MCS was calculated as the sum of the 3 subscores, and the overall score values ranged from 0 to 9, with a higher score indicating more severe disease. Population: The analysis was performed using the intent-to-treat (ITT) population that consisted of all randomized participants who received at least 1 dose of study drug. One subject had missing data at baseline.
  score on a scale
    number analyzed (Participants) | 52 | 50 | 53 | 155
    (all) | 6.5 (1.23) | 6.6 (1.17) | 6.5 (1.51) | 6.5 (1.31)
The 2-component MCS [Mean (Standard Deviation); unit: score on a scale] — The 2-component MCS was used to measure disease activity of ulcerative colitis. It consisted of 2 subscores (rectal bleeding and findings on endoscopy), each of which was rated on a scale from 0 to 3, indicating normal to severe. The 2-component MCS was calculated as the sum of the 2 subscores, and the overall score value ranged from 0 to 6, with a higher score indicating more severe disease. Population: The analysis was performed using the ITT population that consisted of all randomized participants who received at least 1 dose of study drug. One subject had missing data at baseline.
  score on a scale
    number analyzed (Participants) | 52 | 50 | 53 | 155
    (all) | 4.2 (0.75) | 4.2 (0.75) | 4.2 (0.91) | 4.2 (0.80)
Total Mayo Score (TMS) [Mean (Standard Deviation); unit: score on a scale] — The TMS consisted of 4 subscores [stool frequency, rectal bleeding, findings of endoscopy (flexible proctosigmoidoscopy), and Physician's Global Assessment (PGA) score], each of which was rated on a scale from 0 to 3, indicating normal to severe. The TMS was calculated as the sum of the 4 subscores, and the overall score values ranged from 0 to 12, with a higher score indicating more severe disease. Population: The analysis was performed using the ITT population that consisted of all randomized participants who received at least 1 dose of study drug. One subject had missing data at baseline.
  score on a scale
    number analyzed (Participants) | 52 | 50 | 53 | 155
    (all) | 8.8 (1.43) | 8.9 (1.47) | 8.7 (1.72) | 8.8 (1.54)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adapted Mayo Score (MCS) at Week 12
Description: The adapted MCS was used to measure disease activity of ulcerative colitis. It consisted of 3 subscores (stool frequency, rectal bleeding, and findings of endoscopy), each of which was rated on a scale from 0 to 3, indicating normal to severe. The adapted MCS was calculated as the sum of the 3 subscores, and the overall score values ranged from 0 to 9, with a higher score indicating more severe disease. Multiple imputation method was used to handle missing data.
Time Frame: Baseline and Week 12
Population: The analysis was performed using the intent-to-treat (ITT) population that consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
score on a scale | -1.94 [-2.45 to -1.42] | -2.49 [-3.01 to -1.98] | -1.50 [-2.00 to -1.01]
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.0091, ANCOVA — The analysis was performed using an analysis of covariance (ANCOVA) model that incorporated treatment, current oral corticosteroid use, prior exposure to tumor necrosis factor alpha (TNFα) antagonists, and baseline value as covariate; The analysis compared the adapted MCS change from baseline between treatment groups using a 1-sided test at the 0.05 level of significance; Difference in least square mean = -0.99, 90% CI 2-sided [-1.68 to -0.30], Standard Error of Mean 0.42 — Estimated least square mean difference in etrasimod 2 mg from placebo
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.1457, ANCOVA — The analysis was performed using an ANCOVA model that incorporated treatment, current oral corticosteroid use, prior exposure to TNFα antagonists, and baseline value as covariate; [statistical method as in outcome 1, analysis 1]; Difference in least square mean = -0.43, 90% CI 2-sided [-1.11 to 0.24], Standard Error of Mean 0.41 — Estimated least square mean difference in etrasimod 1 mg from placebo

2. Secondary Outcome: Percentage of Participants Who Achieved Endoscopic Improvement at Week 12
Description: For determination of the endoscopic subscore of the MCS, a flexible proctosigmoidoscopy, performed with a videoendoscope following a cleansing prep (oral or rectal cathartic) was performed at screening (within 10 days prior to administration of the first dose of study drug) and the Week 12 visit. This efficacy procedure assessed endoscopic mucosal appearance. The results were rated on a scale from 0 to 3, indicating normal to severe. Endoscopic improvement was defined as Mayo endoscopic subscore (using findings of flexible proctosigmoidoscopy) of ≤1 point. Multiple imputation method was used to handle missing data.
Time Frame: Week 12
Population: The analysis was performed using the ITT population that consisted of all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
percentage of participants | 22.5 | 41.8 | 17.8
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.003, Mantel Haenszel — Mantel-Haenszel (MH) estimated common risk difference adjusted for current oral corticosteroid therapy at baseline and previous exposure to TNFα antagonists; The analysis compared the difference in proportions between treatment groups using a 1-sided test at the 0.05 level of significance; MH estimate for difference in percentage = 24.4, 90% CI 2-sided [9.8 to 39.0], Standard Error of Mean 8.87 — MH estimated difference in etrasimod 2 mg from Placebo
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.3059, Mantel Haenszel — MH estimated common risk difference adjusted for current oral corticosteroid therapy at baseline and previous exposure to TNFα antagonists; [statistical method as in outcome 2, analysis 1]; MH estimate for difference in percentage = 4.1, 90% CI 2-sided [-9.1 to 17.2], Standard Error of Mean 7.98 — MH estimated difference in etrasimod 1 mg from Placebo

3. Secondary Outcome: Change From Baseline in 2-component MCS at Week 12
Description: The 2-component MCS was used to measure disease activity of ulcerative colitis. It consisted of 2 subscores (rectal bleeding and findings on endoscopy), each of which was rated on a scale from 0 to 3, indicating normal to severe. The 2-component MCS was calculated as the sum of the 2 subscores, and the overall score value ranged from 0 to 6, with a higher score indicating more severe disease. Multiple imputation method was used to handle missing data.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
score on a scale | -1.30 [-1.66 to -0.95] | -1.75 [-2.11 to -1.40] | -0.92 [-1.26 to -0.57]
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.0020, ANCOVA — [p-value comment as in outcome 1, analysis 2]; The analysis compared the 2-component MCS change from baseline between treatment groups using a 1-sided test at the 0.05 level of significance; Difference in least square mean = -0.84, 90% CI 2-sided [-1.32 to -0.36], Standard Error of Mean 0.29 — Estimated least square mean difference in etrasimod 2 mg from placebo
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.0858, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 3, analysis 1]; Difference in least square mean = -0.39, 90% CI 2-sided [-0.85 to 0.08], Standard Error of Mean 0.28 — Estimated least square mean difference in etrasimod 1 mg from placebo

4. Secondary Outcome: Change From Baseline in Total Mayo Score (TMS) at Week 12
Description: The TMS was used to measure disease activity of ulcerative colitis. It consisted of 4 subscores [stool frequency, rectal bleeding, findings of endoscopy (flexible proctosigmoidoscopy), and Physician's Global Assessment (PGA) score], each of which was rated on a scale from 0 to 3, indicating normal to severe. The TMS was calculated as the sum of the 4 subscores, and the overall score values ranged from 0 to 12, with a higher score indicating more severe disease. Multiple imputation method was used to handle missing data.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
score on a scale | -2.69 [-3.36 to -2.02] | -3.35 [-4.03 to -2.68] | -2.08 [-2.73 to -1.44]
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.0100, ANCOVA — [p-value comment as in outcome 1, analysis 2]; The analysis compared the TMS change from baseline between treatment groups using a 1-sided test at the 0.05 level of significance; Difference in least square mean = -1.27, 90% CI 2-sided [-2.17 to -0.37], Standard Error of Mean 0.55 — Estimated least square mean difference in etrasimod 2 mg from placebo
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.1277, ANCOVA — [p-value comment as in outcome 1, analysis 2]; [statistical method as in outcome 4, analysis 1]; Difference in least square mean = -0.60, 90% CI 2-sided [-1.48 to 0.27], Standard Error of Mean 0.53 — Estimated least square mean difference in etrasimod 1 mg from placebo

5. Other Pre Specified Outcome: Trichotomous Composite Score of Clinical Remission and Clinical Response at Week 12
Description: The trichotomous composite score of clinical remission and clinical response at Week 12 is an ordinal categorical endpoint with 3 categories (score ranging 0 to 2: score 2 for achieving both clinical remission and clinical response; 1 for only achieving clinical response, and 0 for achieving neither). Multiple imputation method was used to handle missing data.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
score on a scale | 0.60 (0.11) | 0.84 (0.13) | 0.41 (0.09)
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.0071, ANCOVA — The analysis was performed using an ordered logistic regression model with terms for treatment, current oral corticosteroid use, and prior exposure to TNFα antagonists; The analysis compared the odds of achieving higher trichotomous composite score between the groups using 1-sided test at 0.05 level of significance; Odds Ratio (OR) = 2.78, 90% CI 2-sided [1.40 to 5.51]
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.1192, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.61, 90% CI 2-sided [0.83 to 3.14]

6. Other Pre Specified Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 12
Description: A participant was considered to have achieved clinical remission if he/she had: 1) an endoscopy score using flexible proctosigmoidoscopy of 0 or 1 (excluding friability), 2) a rectal bleeding score of 0 or 1, and 3) a stool frequency score of 0 or 1 with a decrease of ≥1 point from baseline. Multiple imputation method was used to handle missing data.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
percentage of participants | 16.0 | 33.0 | 8.1
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.0003, Mantel Haenszel — The analysis was performed using MH method that was adjusted for current oral corticosteroid therapy at baseline and previous exposure to TNFα antagonists; [statistical method as in outcome 2, analysis 1]; MH estimate for difference in percentage = 25.8, 90% CI 2-sided [13.5 to 38.1], Standard Error of Mean 7.47 — MH estimated difference in etrasimod 2 mg from Placebo
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.1360, Mantel Haenszel — [p-value comment as in outcome 6, analysis 1]; [statistical method as in outcome 2, analysis 1]; MH estimate for difference in percentage = 7.1, 90% CI 2-sided [-3.5 to 17.7], Standard Error of Mean 6.46 — MH estimated difference in etrasimod 1 mg from Placebo

7. Other Pre Specified Outcome: Percentage of Participants Who Achieved Clinical Response at Week 12
Description: A participant was considered to have achieved clinical response if he/she met the criteria of clinical remission defined above, or met criteria of clinical response. Clinical response was defined as a decrease in the adapted MCS of ≥ 2 points and a decrease of ≥ 30% with either a decrease of rectal bleeding of ≥ 1 or rectal bleeding score of 0 or 1.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 52 | 50 | 54
percentage of participants | 43.7 | 50.6 | 32.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; The primary comparison in the study was between etrasimod 2 mg versus placebo; Test type: Superiority; p = 0.0282, Mantel Haenszel — [p-value comment as in outcome 6, analysis 1]; [statistical method as in outcome 2, analysis 1]; MH estimate for difference in percentage = 18.9, 90% CI 2-sided [2.6 to 35.3], Standard Error of Mean 9.92 — MH estimated difference in etrasimod 2 mg from Placebo
Statistical Analysis 2: Comparison: Etrasimod 1 mg vs Placebo; Test type: Superiority; p = 0.1309, Mantel Haenszel — [p-value comment as in outcome 6, analysis 1]; [statistical method as in outcome 2, analysis 1]; MH estimate for difference in percentage = 11.4, 90% CI 2-sided [-5.3 to 28.1], Standard Error of Mean 10.14 — MH estimated difference in etrasimod 1 mg from Placebo

ADVERSE EVENTS:
Time Frame: Up to approximately 16 weeks i.e. from the time of administration of the first dose of study drug up to 30 days after the administration of the last dose of study drug.
Description: Treatment-Emergent Adverse Event (TEAE) were collected during the study.
Arm/Group | Etrasimod 1 mg | Etrasimod 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 0/54
Serious Adverse Events (participants affected / at risk) | 3/52 | 0/50 | 6/54
Other Adverse Events (participants affected / at risk) | 11/52 | 11/50 | 9/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 1 mg (N=52) | Etrasimod 2 mg (N=50) | Placebo (N=54)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 1 mg (N=52) | Etrasimod 2 mg (N=50) | Placebo (N=54)
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2
Colitis ulcerative (Gastrointestinal disorders) | 3 | 2 | 1
Headache (Nervous system disorders) | 0 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT02447302/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT02447302/SAP_001.pdf